CLINICAL TRIAL: NCT02846064
Title: Development of Ovarian Tissue Autograft in Order to Restore Ovarian Function
Acronym: DATOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: CHU de Reims (Other); University Hospital, Marseille (Other); Nantes University Hospital (Other); University Hospital, Lille (Other); Central Hospital, Nancy, France (Other); University Hospital, Toulouse (Other); University Hospital, Grenoble (Other); University Hospital, Bordeaux (Other); CMCO SIHCUS, Schiltingheim (Other); University Hospital, Rouen (Other); University Hospital, Limoges (Other); University Hospital, Angers (Other Government); Centre Hospitalier Universitaire de Nice (Other); Tenon Hospital, Paris (Other); Poissy-Saint Germain Hospital (Other); Hôpital Jean Verdier (Other); University Hospital, Clermont-Ferrand (Other); Hopital Antoine Beclere (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2012/143
Record Dates: First submitted 2013-10-25; First posted 2016-07-27 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Function Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ovarian tissue cryopreservation (Other)
  Interventions: Procedure: Autograft of cryopreserved ovarian tissue

INTERVENTIONS:
Procedure: Autograft of cryopreserved ovarian tissue — Orthotopic transplantation

SUMMARY:
Ovarian cryopreservation is one of the available option for preserving fertility prior to potentially sterilizing treatments. In the absence of other techniques such as in vitro folliculogenesis or injection of isolated ovarian follicles, this tissue can only be re-used by autograft. In France, the first live birth after orthotopic ovarian transplantation, was obtained by Roux et al. in 2009. This clinical trial aims to collect data on the efficiency of the graft in terms of restoration of ovarian function and live births. It will also allow us to carry out the patient follow-up after ovarian tissue cryopreservation and after autograft when achieved. In cases of neoplastic malignancies, minimal residual disease detection will be performed on ovarian tissue, to avoid any risk of cancer re-seeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Ovarian tissue cryopreservation
* Premature ovarian failure
* Patients cured of their primary disease
* Women between 18 and 43 years of age
* Patients who have already benefited from ovarian tissue autograft

Exclusion Criteria:

* Patients under trusteeship
* Patients placed in receivers
* Patients under the protection of a conservator

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Restoration of ovarian function by using autograft | 2 years

SECONDARY OUTCOMES:
Number of live births after ovarian tissue autograft | 5 years
Number of complications that could result from a surgery with anesthesia or depending on graft quality | 5 years
Number of graft recovery | 5 years
Number of residual disease development. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besancon, Besançon, France

REFERENCES:
- [Background] Roux C, Amiot C, Agnani G, Aubard Y, Rohrlich PS, Piver P. Live birth after ovarian tissue autograft in a patient with sickle cell disease treated by allogeneic bone marrow transplantation. Fertil Steril. 2010 May 1;93(7):2413.e15-9. doi: 10.1016/j.fertnstert.2009.12.022. Epub 2010 Feb 1. PMID 20117783
- [Background] Amiot C, Angelot-Delettre F, Zver T, Alvergnas-Vieille M, Saas P, Garnache-Ottou F, Roux C. Minimal residual disease detection of leukemic cells in ovarian cortex by eight-color flow cytometry. Hum Reprod. 2013 Aug;28(8):2157-67. doi: 10.1093/humrep/det126. Epub 2013 Apr 30. PMID 23633552
- [Background] Fauque P, Ben Amor A, Joanne C, Agnani G, Bresson JL, Roux C. Use of trypan blue staining to assess the quality of ovarian cryopreservation. Fertil Steril. 2007 May;87(5):1200-7. doi: 10.1016/j.fertnstert.2006.08.115. Epub 2007 Feb 20. PMID 17307173
- [Background] Pretalli JB, Frontczak Franck S, Pazart L, Roux C, Amiot C; DATOR Group. Development of Ovarian Tissue Autograft to Restore Ovarian Function: Protocol for a French Multicenter Cohort Study. JMIR Res Protoc. 2019 Sep 30;8(9):e12944. doi: 10.2196/12944. PMID 31573931